CLINICAL TRIAL: NCT03356028
Title: Pedopsychiatric and Multidisciplinary Research (Public Health, Psychodynamics, Neuroscience and Human and Social Sciences) Devoted to Children Exposed to the Attack in Nice on July 14, 2016
Brief Title: Pedopsychiatric and Multidisciplinary Research Devoted to Children Exposed to the Attack in Nice on July 14, 2016
Acronym: Program14-7
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-HPNCL-03
Record Dates: First submitted 2017-11-09; First posted 2017-11-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Psychiatric Disorder; Trauma, Psychological
Keywords: Trauma; Psychiatric Disorder; mass trauma
MeSH Terms: conditions — Mental Disorders; Psychological Trauma; Wounds and Injuries | interventions — Adolescent Psychiatry

STUDY DESIGN:
Intervention Model Description: Interventional research involving the category 2 human person at minimal risk and constraint, excluding health product, multicentre
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- impacted by the attack of 14 July 2016 (Other): characterize the psycho-social factors of risk and / or protection interfering in the children's future with questionnaire following the mass trauma of 14 July 2016 in Nice on a sample of exposed pediatric population
  Interventions: Behavioral: Child and adolescent psychiatry and Epidemiology; Other: salivary biological collection; Behavioral: qualitative analysis of the discourse; Behavioral: Parenthood; Behavioral: Cognitive alterations; Behavioral: Impact on schooling; Behavioral: Sleep disorders and associated somatizations
- control group (Other): characterize the psycho-social factors of risk and / or protection interfering in the children's future with questionnaire of children controls
  Interventions: Behavioral: Child and adolescent psychiatry and Epidemiology

INTERVENTIONS:
Behavioral: Child and adolescent psychiatry and Epidemiology — psychosocial risk assessment questionnaire, structured diagnostic interview, pedopsychiatric questionnaire
Other: salivary biological collection — Saliva sampling will be done using a specific kit
  Arms: impacted by the attack of 14 July 2016
Behavioral: qualitative analysis of the discourse — two semi-structured interviews, the first with the teenager alone, the second with the lone parents
  Arms: impacted by the attack of 14 July 2016
Behavioral: Parenthood — Parenting Sense of Competence (PSOC) questionnaires completed online.Two visits will be realized: a first in the month preceding the start of the trial and a second in the month following the end of the trial
  Arms: impacted by the attack of 14 July 2016
Behavioral: Cognitive alterations — Episodic memory will be assessed using Grober and Buschke. The evaluation of the cognitive alterations will include two stages: a first in the month preceding the start of the trial and a second in the month following the end of the trial. For child and parents
  Arms: impacted by the attack of 14 July 2016
Behavioral: Impact on schooling — collect of several data about the number of absences of the child, the number of exclusions and hours of detention of the child, as well as the school reports of the child
  Arms: impacted by the attack of 14 July 2016
Behavioral: Sleep disorders and associated somatizations — Evaluation of sleep disorders and associated somatizations by connected watche and sleep questionnaire
  Arms: impacted by the attack of 14 July 2016

SUMMARY:
On July 14, 2016, in Nice, children and their families were attacked by the organization "EI". In Nice, 86 deaths, including 10 children, the youngest at 4, were recorded. A number of children, still difficult to assess exactly but over 100, was bereaved.

After a traumatic event, multiple clinical consequences may appear in children. Among these consequences, the most common is Post-Traumatic Stress Disorder (PTSD). The aim of the study is to characterize the psycho-social factors of risk and / or protection interfering in the children's future, following the mass trauma of 14 July 2016 in Nice on a sample of pediatric population exposed in comparison of children controls.

Ancillary study, entilted "The Physalis Child", prospectively observe the presence or not of non-psychotic acousto-verbal hallucinations (AVH) in the population with PTSD from the "Program 14-7". The main objective of this ancillary study will be to identify factors of social and emotional cognition linked to the presence of non-psychotic HAV within the cohort of children exposed to the mass trauma of July 14, 2016 in Nice but also to any type of individual trauma.

Ancillary study, entilted "trail of the 14 July attack", prospectively observe the risk of traumatic reactivation.

DETAILED DESCRIPTION:
On July 14, 2016, in Nice, children and their families were attacked by the organization "EI". This is the second time in our country that children are victims of this organization after the attack on the school Ozar Hotarah in March 2012 in Toulouse where four children were killed "touching end".

In Nice, 86 deaths, including 10 children, the youngest at 4, were recorded. A number of children, still difficult to assess exactly but over 100, was bereaved.

After a traumatic event, multiple clinical consequences may appear in children. Among these consequences, the most common is Post-Traumatic Stress Disorder (PTSD). This pathology includes 4 main symptoms: the reviviscences of the event, avoidance behaviors, alterations of cognition and mood and neurovegetative overactivation. In addition, PTSD contributes to the development of many other mental disorders. It is estimated that 75% of adolescents or children having a comorbid disorder with PTSD. In the literature, the main comorbidities identified in pediatric populations are: anxiety disorders, Attention Deficit Hyperactivity Disorder (ADHD) and depression. There is no recommendation as to the therapeutics to be used in psychotraumatism in pediatric population. Epidemiological studies conducted on the consequences of trauma reveal a high variability in the development of psychopathologies. 6 to 20% of exposed children would develop PTSD after a potentially traumatic situation. Several factors can explain the heterogeneity of the results, including the age, the type of trauma experienced, the violence suffered during this trauma. In Nice, to date, more than 2200 children have consulted: 700 children between July 14 and July 28, 2016, 1100 children were seen between August and December, and about 400 since the creation of the Post Traumatic Pediatric Intersectoral Assessment Center (CE2P), in January 2017. The aim of the study is to characterize the psycho-social factors of risk and / or protection interfering in the children's future, following the mass trauma of 14 July 2016 in Nice on a sample of pediatric population exposed in comparison of children controls.

Non-psychotic hallucinations represent a significant symptomatology in child psychiatry (1) and remain clinical question. The results of our previous study "the physalis child" showed a significant correlation between the persistence of non-psychotic acousto-verbal hallucinations (AVH) and the presence of negative emotions, linked to post traumatic stress disorder (PTSD). It seems important to understand the link between trauma and the presence of non-psychotic AVH in children as the literature shows the risk of progression to psychosis when these AVH persist.The interest of the ancllary study of "the physalis child" would be to prospectively observe the presence or not of non-psychotic AVH in the population with PTSD from the "Program 14-7". The question would then be: "Why in two subjects diagnosed with PTSD, one has non-psychotic HAV and the other does not?" The main objective of this ancillary study will be to identify factors of social and emotional cognition linked to the presence of non-psychotic HAV within the cohort of children exposed to the mass trauma of July 14, 2016 in Nice but also to any type of individual trauma.

The impending opening of the trial of the 14 July attack, the conduct and the media coverage associated with the trial are all factors that could be distressing for the children and families exposed to the attack in Nice. Re-exposure to testimonials and certain images can increase the risk of traumatic reactivation with a return of suppressed fears and the symptoms associated. Some factors have been identified as protective: social and family support, cognitive functioning, the presence of residual symptoms or the quality of sleep.

Therefore, an assessment of these factors before and after the opening of the trial would identify children and families with traumatic reactivation, as well as identify protective or risk factors for relapse of traumatic symptoms

ELIGIBILITY:
Inclusion Criteria:

* Children and / or young adults who have consulted at the pediatric consultation center of the CHU Lenval or who are listed in the ORSAN "organization of the health system response in exceptional health situations" file or who have made an appointment following the call by press;
* Children and / or young adults under 18 at the time of the Nice attack of 14/07/2016.
* Affiliated to a social security scheme;
* Having a good command of the French language (French);
* Children whose parents have accepted participation in the study (collection of informed consents).

Non inclusion:

* Children and / or young adults with average intellectual disability (Intelligence Quotient IQ less than 50);
* Person deprived of liberty by judicial or administrative decision;
* Person subject to an exclusion period for another search.

Exclusion Criteria:

* a simple request from the child / adolescent and / or young adults or their parents (interruption of participation or withdrawal of consent);
* failure to comply with the instructions defined and exposed at the time of inclusion.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 728 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2044-12 (Estimated); Study Completion 2044-12 (Estimated)

PRIMARY OUTCOMES:
psychosocial risk assessment questionnaire after 2 year | Difference between baseline and after 2 year
  Completion of the psychosocial risk assessment questionnaire

SECONDARY OUTCOMES:
psychosocial risk assessment questionnaire after 5 year | Difference between baseline and after 5 year
  Completion of the psychosocial risk assessment questionnaire
psychosocial risk assessment questionnaire after 10 year | Difference between baseline and after 10 year
  Completion of the psychosocial risk assessment questionnaire
psychosocial risk assessment questionnaire after 15 year | Difference between baseline and after 15 year
  Completion of the psychosocial risk assessment questionnaire
psychosocial risk assessment questionnaire after 20 year | Difference between baseline and after 20 year
  Completion of the psychosocial risk assessment questionnaire
psychosocial risk assessment questionnaire after 25 year | Difference between baseline and after 25 year
  Completion of the psychosocial risk assessment questionnaire
Structured diagnostic interview MINI (Mini International Neuropsychiatric Interview) after 2 year | Difference between baseline and after 2 year
  Completion of the MINI questionnaire
Structured diagnostic interview MINI (Mini International Neuropsychiatric Interview) after 5 year | Difference between baseline and after 5 year
  Completion of the MINI questionnaire
Structured diagnostic interview MINI (Mini International Neuropsychiatric Interview) after 10 year | Difference between baseline and after 10 year
  Completion of the MINI questionnaire
Structured diagnostic interview MINI (Mini International Neuropsychiatric Interview) after 15 year | Difference between baseline and after 15 year
  Completion of the MINI questionnaire
Structured diagnostic interview MINI (Mini International Neuropsychiatric Interview) after 20 year | Difference between baseline and after 20 year
  Completion of the MINI questionnaire
Structured diagnostic interview MINI (Mini International Neuropsychiatric Interview) after 25 year | Difference between baseline and after 25 year
  Completion of the MINI questionnaire
Overall assessment of the individual CGI-S (Clinical Global Impression - Severity) after 2 year | Difference between baseline and after 2 year
  Completion of the CGI-S
Overall assessment of the individual CGI-S (Clinical Global Impression - Severity) after 5 year | Difference between baseline and after 5 year
  Completion of the CGI-S
Overall assessment of the individual CGI-S (Clinical Global Impression - Severity) after 10 year | Difference between baseline and after 10 year
  Completion of the CGI-S
Overall assessment of the individual CGI-S (Clinical Global Impression - Severity) after 15 year | Difference between baseline and after 15 year
  Completion of the CGI-S
Overall assessment of the individual CGI-S (Clinical Global Impression - Severity) after 20 year | Difference between baseline and after 20 year
  Completion of the CGI-S
Overall assessment of the individual CGI-S (Clinical Global Impression - Severity) after 25 year | Difference between baseline and after 25 year
  Completion of the CGI-S
General operation CGA-S (Children's Global Assessment Scale) after 2 year | Difference between baseline and after 2 year
  Completion of the CGA-S
General operation CGA-S (Children's Global Assessment Scale) after 5 year | Difference between baseline and after 5 year
  Completion of the CGA-S
General operation CGA-S (Children's Global Assessment Scale) after 10 year | Difference between baseline and after 10 year
  Completion of the CGA-S
General operation CGA-S (Children's Global Assessment Scale) after 15 year | Difference between baseline and after 15 year
  Completion of the CGA-S
General operation CGA-S (Children's Global Assessment Scale) after 20 year | Difference between baseline and after 20 year
  Completion of the CGA-S
General operation CGA-S (Children's Global Assessment Scale) after 25 year | Difference between baseline and after 25 year
  Completion of the CGA-S
identify factors of social cognition linked to the presence of non-psychotic acousto-verbal hallucinations (AVH) | at baseline
  completion of the NEPSY II for a complete neuropsychological assessment
identify factors of emotional cognition linked to the presence of non-psychotic AVH | at baseline
  completion of the EED IV , French version of the Differential Emotions Scale IV (DES-IV
identify the factors of persistence of AVH | after 6 months, 1 year and 2 year from baseline
  complete neuropsychological assessment
impact of trial of the attack July 14th on Parenthood | baseline and month9
  Parenthood assessment will be offered to parents of children included in the arm "impacted by attack" The Parenting Sense of Competence (PSOC) questionnaire is a widely used scale to assess and measure parenting abilities perceived by parents with two subscales: competence/knowledge and appreciation/comfort.
  The PSOC is a scale with a score ranging from 17 to 102. The higher the score, the more the parent feels a sense of high parenting competence. To demonstrate a minimum difference of 20 points on this questionnaire before and after the trial, with a standard deviation of 20, the number of participants required is 44
  Two visits will be realized: a first in the month preceding the start of the trial (baseline) and a second in the month following the end of the trial.
impact of trial of the attack July 14th on Cognitive alterations | baseline and month 6
  Evaluation of cognitive alterations, in particular memory disorders and executive functions, will be aimed at children aged 0 to 6 at the time of the July 14, 2016 attack Episodic memory will be assessed using Grober and Buschke (Grober and Buschke, 1988). This test includes 16 items to memorize belonging to 16 different semantic categories. The duration of this test is approximately 20 minutes. This test starts with a control phase of the semantic encoding of words with an immediate cued recall, 3 free and cued recall phases with a 20-second interferential task, a recognition phase and finally a free and deferred cued recall phase to test learning.
  Previous studies using this test show a mean difference of 2 points between the control groups and the experimental groups.
  The evaluation of the cognitive alterations will include two stages: a first in the month preceding the start of the trial (baseline) and a second in the month following the end of the trial
impact of trial of the attack July 14th on schooling | 2 years from baseline
  Evaluation of the impact of schooling will focus on middle and high school students, using Pronote software and included in the arm "impacted by attack" .
  In order to test the impact of the trial on children's education, several data will be requested from parents. Using the Pronote software, they will be able to communicate to us the number of absences of the child, the number of exclusions and hours of detention of the child, as well as the school reports of the child to obtain the effective grades of children and adolescents. This data will be collected for the 2021-2022 school year (3 terms of the previous school year) and for the 2022-2023 school year (3 terms of the current year).
impact of trial of the attack July 14th on Sleep disorders and associated somatizations | baseline and month 6
  Evaluation of sleep disorders and associated somatizations will be offered to adolescents in the "14-7" cohort, are children aged 7 to 12 at the time of the attack.
  The screening scale for sleep disorders in children aged 4 to 16 years by Bruni et al. 1996 . This questionnaire includes an overall sleep quality score, but also sub-indices evaluating insomnia, parasomnia, respiratory problems, non-restorative sleep and excessive daytime sleepiness. The threshold score is 39 and an average score around 25 for the control population.
  This questionnaire will be carried out during the month preceding the opening of the trial (baseline), then every month, until the end of the trial.
  From baseline to the end of trial, participants will receive a connected watches to continuously record sleep quality and daytime activity.
  A questionnaire on Post Traumatic Stress Disorder (PTSD) symptoms will also be completed by the participants at baseline and at the end of trial.

CONTACTS AND LOCATIONS:
Overall Officials: Florence ASKENAZY, MD, Principal Investigator — Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (1):
- Hôpitaux pédiatriques de Nice CHU-Lenval, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dumas LE, Askenazy F, Fernandez A. Relationships between markers of emotional and social cognition and acoustic-verbal hallucinations in children and adolescents with post-traumatic stress disorder (PTSD). PLoS One. 2025 Sep 23;20(9):e0332910. doi: 10.1371/journal.pone.0332910. eCollection 2025. PMID 40986567
- [Derived] Dumas LE, Fernandez A, Auby P, Askenazy F. Relationship between social cognition and emotional markers and acoustic-verbal hallucination in youth with post-traumatic stress disorder: Protocol for a prospective, 2-year, longitudinal case-control study. PLoS One. 2024 Jul 2;19(7):e0306338. doi: 10.1371/journal.pone.0306338. eCollection 2024. PMID 38954699
- [Derived] Gindt M, Thummler S, Soubelet A, Guenole F, Battista M, Askenazy F. Methodology of "14-7" Program: A Longitudinal Follow-Up Study of the Pediatric Population and Their Families Exposed to the Terrorist Attack of Nice on July 14th, 2016. Front Psychiatry. 2019 Sep 12;10:629. doi: 10.3389/fpsyt.2019.00629. eCollection 2019. PMID 31572232